CLINICAL TRIAL: NCT00547027
Title: Promoting Physical Activity Among Patients With Type 2 Diabetes in a Community-Based Clinic
Brief Title: Promoting Physical Activity Among Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Florida State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG 017294
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes; Physical Activity
Keywords: diabetes; physical activity; print-based intervention; tailored intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: print-based physical activity intervention — individually-based, print-based physical activity intervention
Behavioral: usual care — print-based materials of nutritional information

SUMMARY:
The purpose of this study is to determine the effects of a tailored, print-based physical activity intervention for patients diagnosed with type 2 diabetes.

DETAILED DESCRIPTION:
Given the growing rates of type 2 diabetes and the documented benefits of physical activity in the treatment of this illness, further research is needed to examine methods of targeting this patient group to achieve improvements in physical activity behavior. The primary aim of this planning grant is to implement a pilot study examining the feasibility and efficacy of an individually-targeted, theoretically-based physical activity intervention for patients with type 2 diabetes. The physical activity intervention is compared to usual care, and the primary outcome is weekly physical activity at a one-month follow-up. These pilot data would demonstrate the feasibility of partnering with a community agency for participant recruitment and program implementation, as well as the potential efficacy of this intervention to promote physical activity in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* adults diagnosed with type 2 diabetes
* current patients referred to diabetes center

Exclusion Criteria:

* medical contra-indication to moderate-intensity physical activity

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2006-04; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
weekly physical activity | one month

SECONDARY OUTCOMES:
physical activity stage of change | one month

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Dutton, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States